CLINICAL TRIAL: NCT05226117
Title: SURE-01_An Open Label, Single-arm, Phase 2 Study of Neoadjuvant Sacituzumab Govitecan, Before Radical Cystectomy, for Patients With Muscleinvasive Bladder Cancer Who Cannot Receive or Refuse Cisplatin-based Chemotherapy
Brief Title: Sacituzumab Govitecan, Preceding Radical Cystectomy, in Treating Patients With Muscle-invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: High Research (Other)
Responsible Party: Principal Investigator, Prof. Andrea Necchi, Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURE-01
Record Dates: First submitted 2022-01-08; First posted 2022-02-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Patients with muscle-invasive urothelial carcinoma of the bladder, who are suited for and accept radical cystectomy (RC)
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — Sacituzumab govitecan is a humanized monoclonal antibody (mAb) with a hydrolyzable linker through which SN-38 is conjugated to the humanized mAb hRS7 IgG1κ to enhance the delivery of SN-38 to Trop-2- expressing tumors while reducing systemic toxicity. SN-38 is the active metabolite of irinotecan. Sacituzumab govitecan is administered at 7.5 mg/kg as an IV infusion on days 1 and 8 of a 21- day cycle till progression, toxicity or withdrawal of consent

SUMMARY:
SURE-01 is a neoadjuvant phase 2, open-label, non-randomized, singlecohort study in patients with urothelial carcinoma of the bladder. Patients will be consecutively enrolled and treated. The primary objective of the study is to assess whether sacituzumab govitecan results in pathological complete response (in patients with Muscle-invasive Bladder Cancer who cannot receive or refuse cisplatin-based chemotherapy). Secondary objectives were to evaluate the radiological response of those patients with measurable disease; to evaluate the surgical and medical safety of neoadjuvant therapy; to assess survival outcomes (event-free survival and overall survival).

DETAILED DESCRIPTION:
SURE-01 is a neoadjuvant phase 2, open-label, non-randomized, singlecohort study in patients with urothelial carcinoma of the bladder. Patients will be consecutively enrolled and treated. The primary objective of the study is to assess whether sacituzumab govitecan results in pathological complete response (in patients with Muscle-invasive Bladder Cancer who cannot receive or refuse cisplatin-based chemotherapy). Secondary objectives were to evaluate the radiological response of those patients with measurable disease; to evaluate the surgical and medical safety of neoadjuvant therapy; to assess survival outcomes (event-free survival and overall survival).

The general framework of the study will be as follows:

A transurethral resection of the bladder tumor (TURBT) for biopsy, histological characterization, and local staging will be executed first, according to the guidelines. With the aim to improve the sensitivity of computed tomography (CT) scan in assessing pelvic lymph-nodes and better assess the local extent of bladder tumor, CT scan, 18F-fluorodeoxyglucose positron emission tomography (18FDG-PET)/CT scan, and multiparametric bladder magnetic resonance imaging (mpMRI) will be done during screening and before cystectomy to stage and evaluate response.

* Eligible patients will receive neoadjuvant treatment: 7.5 mg/kg sacituzumab govitecan IV, on days 1, 8, of each 21 day cycle.
* A total of 4 cycles is planned before surgery. Surgery will be planned at the time of study inclusion to be done within 4 weeks of the last dose of study drug. After surgery patients will be managed according to local guidelines which mirror the current EAU guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects, >18 years of age, able to understand and give written informed consent
2. Histopathologically confirmed urothelial carcinoma. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) transitional cell pattern.
3. Fit and planned for RC (according to local guidelines).
4. ECOG performance status score of 0 or 1
5. Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (Hemoglobin ≥ 9 g/dL, absolute neutrophil count≥ 1,500/ mm3, and Platelets ≥ 100,000/ μL)
6. Adequate hepatic function (Bilirubin ≤ 1.5 IULN, aspartate aminotransferase and alanine aminotransferase≤ 2.5 x IULN or ≤ 5 x IULN if known liver metastases and serum albumin >3 g/dl)
7. Creatinine clearance ≥30 mL/min as assessed by the Cockcroft-Gault equation
8. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication, and must not be lactating. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
9. Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >2 years
10. Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of study therapy.
11. Clinical stage defining clinical T2-T4N0M0 disease by CT (or MRI) + PET/CT (within 4 weeks of randomization by RECIST v1.1).
12. The patient accepts to undergo radical cystectomy.
13. Ineligibility to receive cisplatin-based neoadjuvant chemotherapy based on Galsky's criteria OR refusal to receive neoadjuvant cisplatin-based chemotherapy.

Exclusion Criteria:

1. Have received prior systemic anti-cancer therapy including investigational agents and immunotherapy.
2. Have received prior radiotherapy on the bladder tumor.
3. Refusal to undergo RC.
4. Are currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
5. Have a known additional malignancy that is progressing or has required active treatment within the past 3 years.
6. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer defined as follows are not excluded; Stage T1c or T2a with a Gleason score ≤ 6 and prostatic-specific antigen (PSA) < 10 ng/mL either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study allocation. Women who are pregnant or lactating
7. Have severe hypersensitivity (≥Grade 3) to sacituzumab govitecan and/or any of its excipients.
8. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
9. Have nephrostomy, central venous catheters, any other types of catheters that could make the patient at higher risk of developing severe infectious complications during treatment with sacituzumab govitecan.
10. Have ≥3 risk factors for the development of febrile neutropenia according to the ASCO guidelines (Smith et al, J Clin Oncol. 2015;33:3199-3212). These risk factors are the following: Age >65 years, advanced disease, Previous chemotherapy or radiation therapy, Preexisting neutropenia or bone marrow involvement with tumor, infection, Open wounds or recent surgery, Poor performance status or poor nutritional status, Poor renal function, Liver dysfunction, most notably elevated bilirubin, Cardiovascular disease, Multiple comorbid conditions, HIV infection.
11. Have a history of inflammatory bowel disease, ulcerative colitis, or any other pre-existing inflammatory or autoimmune disease that could make the patient at higher risk of developing severe diarrhea or related complications.
12. Have active cardiac disease, defined as:

    * Myocardial infarction or unstable angina pectoris within 6 months of C1D1
    * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation
    * NYHA Class III or greater congestive heart failure or left ventricular ejection fraction of < 40%
13. Have a known history of HIV-1/2.
14. Have active Hepatitis B virus (HBV) or Hepatitis C Virus (HCV). In subjects with a history of HBV or HCV, subjects with detectable viral loads will be excluded.
15. Have other concurrent medical or psychiatric conditions that, in the Investigator's opinion may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | After the last cycle of the investigational drug (each cycle is 21 days)
  Pathological complete response will be defined as the absence of any residual viable tumor in the radical cystectomy specimen. Two independent pathologists, blinded to the study findings, with >10 years of experience in genitourinary tumors will independently evaluate the response. The pathological response assessment will be centralized and externally reviewed at San Raffaele Hospital and Scientific Institute, Milan, Italy.

SECONDARY OUTCOMES:
Radiological response | At baseline and within 2 weeks after the last cycle of the investigational drug (each cycle is 21 days)
  Radiological response on those patients with measurable disease will be evaluated by CT scans with contrast of chest/abdomen/pelvis, with a whole body fluorodeoxyglucose positron emission tomography, and with a multiparametric MRI of the bladder. RECIST v1.1 criteria will be used to assess patient the radiological response to treatment.
Perioperative outcomes | During hospitalization for the surgery and at 30- and 90-day after surgery
  Perioperative outcomes will be systematically and prospectively collected at surgery and during hospitalization, as well as at 30- and 90-day after surgery during patient interviews done by medical doctors and according to the EAU guidelines on reporting and grading of complications, as previously reported by our group within the PURE-01 study (Briganti A, et al. Eur Urol 2020;77:576-580).
Survival outcomes | At the end of study, an average 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No